CLINICAL TRIAL: NCT03400566
Title: Effects of Congruent and In-congruent Experiential Learning on Intake of a Novel Vegetable in Preschool Children
Brief Title: Effects of Experiential Learning on Vegetable Intake in Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Economic and Social Research Council, United Kingdom (Other); Purely Nutrition Ltd (Unknown)
Responsible Party: Principal Investigator, Chandani Nekitsing, Postgraduate Research Student, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ULeeds
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Food Habits; Food Preferences; Health Behavior; Diet Habit; Child Behavior
MeSH Terms: conditions — Feeding Behavior; Food Preferences; Health Behavior; Child Behavior | interventions — Narrative Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Narrative (target) (Experimental): Children will receive the story featuring the target vegetable and NO sensory experience.
  Interventions: Behavioral: Narrative
- Narrative+ experiential (target) (Experimental): Children will receive the story featuring the target vegetable and experiential learning with the target vegetable.
  Interventions: Behavioral: Narrative; Behavioral: Experiential
- Narrative (control) (Active Comparator): Children will receive the story featuring the control vegetable and NO sensory experience.
  Interventions: Behavioral: Narrative
- Narrative+ experiential (control) (Active Comparator): Children will receive the story featuring the control vegetable and experiential learning with the control vegetable.
  Interventions: Behavioral: Narrative; Behavioral: Experiential

INTERVENTIONS:
Behavioral: Narrative — Children will be read a story book featuring vegetables for a minimum of 7 times (including twice during the familiarization phase).
Behavioral: Experiential — Children will receive hands on experience with the vegetable. They will get to listen, see, feel, touch and smell the actual vegetable during the two familiarization phases.
  Arms: Narrative+ experiential (control); Narrative+ experiential (target)

SUMMARY:
The aim of this cluster randomized control trial is to test the efficacy of providing experience of a target novel vegetable within the context of an interactive story time to increase intake of the target novel vegetable in preschool aged children (aged 2-5 years).

DETAILED DESCRIPTION:
The aim of this study is to test the efficacy of providing experience of a target novel vegetable within the context of an interactive story time to increase intake of the target novel vegetable in preschool aged children (aged 2-5 years). In particular, the study will assess whether these strategies are effective to encourage intake of an unfamiliar vegetable in children who are fussy eaters.

There are two manipulations in this study - the provision of a story which features either a target vegetable (celeriac) or a control vegetable (carrot) and the presence of experiential learning (smelling, touching, looking at the vegetable) with either the target vegetable or the control vegetable.

Baseline consumption and familiarity of the target veg will be assessed for all children, before the intervention. The intervention consists of two familiarization trials, and 2-weeks of access to a story book featuring vegetables. Following the final familiarization trial, consumption and familiarity will be assessed again. Each familiarization trial consists of a story in class, and depending on condition, an experiential learning episode in class. During the 2 week interval between familiarization sessions nurseries will be requested to ready the story book 5 times in the preschool room (at times convenient to them).

Participants will be cluster randomized into 4 groups (2X2 between subjects design): 1) target vegetable narrative, 2) target vegetable narrative + experiential, 3) control vegetable narrative 4) control vegetable narrative + experiential

Child's food fussiness data will be collected by parents using the Food Fussiness sub scale of the Child Eating Behaviour Questionnaire. Their usual consumption of the target vegetable will also be measured using parent report.

Nursery staff will be requested to provide feedback to evaluate intervention feasibility, barriers and efficacy.

It is predicted that children's intake of the novel vegetable will vary by intervention. The primary hypothesis to be tested is that providing experience of a target novel vegetable within the context of an interactive story time will encourage preschoolers to taste, try and eat the target vegetable.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 5 years old
* Attends nursery on selected test day

Exclusion Criteria:

* Relevant food allergy (celeriac / celery)
* Medical condition which would prevent them from eating the test vegetable

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 337 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Change in intake of the target vegetable | Change in intake of the target vegetable from Baseline to day 14
  Intake of the novel vegetable will be measured at baseline (day 1) and post intervention (day 14). Intake of the novel vegetable will be measured individually and objectively using weight in grams. Change in intake will be calculated by subtraction of baseline intake from post intervention intake.

SECONDARY OUTCOMES:
Knowledge of the target vegetable | Knowledge of the target vegetable at day 14 (post intervention)
  Children's knowledge of the target vegetable will be assessed at baseline (day 1) and post intervention (day 14). Children will be asked to name the photo card featuring the target vegetable.

CONTACTS AND LOCATIONS:
Overall Officials: Chandani Nekitsing, MSc, Principal Investigator — University of Leeds
Locations (1):
- School of Psychology, University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nekitsing C, Blundell-Birtill P, Cockroft JE, Fildes A, Hetherington MM. Increasing Intake of an Unfamiliar Vegetable in Preschool Children Through Learning Using Storybooks and Sensory Play: A Cluster Randomized Trial. J Acad Nutr Diet. 2019 Dec;119(12):2014-2027. doi: 10.1016/j.jand.2019.05.017. Epub 2019 Aug 1. PMID 31378648
- [Derived] Nekitsing C, Blundell-Birtill P, Cockroft JE, Hetherington MM. Taste Exposure Increases Intake and Nutrition Education Increases Willingness to Try an Unfamiliar Vegetable in Preschool Children: A Cluster Randomized Trial. J Acad Nutr Diet. 2019 Dec;119(12):2004-2013. doi: 10.1016/j.jand.2019.05.012. Epub 2019 Aug 1. PMID 31378647